CLINICAL TRIAL: NCT01616797
Title: A Novel Neurobehavioral Intervention for Emotion Regulation in Anxiety and Depression
Brief Title: A Novel Neurobehavioral Intervention for Emotion Regulation in Anxiety and Depression Across the Lifespan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Etkin, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-24813
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Depression, Anxiety; Cognitive Training; Emotion Training; Emotion Regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized intervention (Experimental): Participants will be asked to visit a customized website and engage in computerized exercises. Cognitive and emotion training games.
  Interventions: Behavioral: Computerized neurobehavioral intervention
- Control (Sham Comparator): Participants will be asked to visit a customized website and engage in computerized games.
  Interventions: Behavioral: Computerized neurobehavioral intervention

INTERVENTIONS:
Behavioral: Computerized neurobehavioral intervention — Participants will complete the intervention by logging into a secure online website and complete computerized neurobehavioral tasks. Tasks will train the following - cognitive control, working memory and task shifting with two different tasks that engage these skills and positivity biases.

SUMMARY:
The research proposes to use an innovative solution to shape brain circuits that support executive function and emotion reactivity -using targeted neurobehavioral intervention.

DETAILED DESCRIPTION:
Participants will be recruited locally in the San Francisco Bay area with certain symptoms of anxiety and depression. They will complete a clinical assessment and then take part in a cognitive-emotion training delivered online.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression on the SCID, a total Ham-D≥16 and Ham-D anxiety/somatization subscale ≥ 7.

Exclusion Criteria:

* Current medication for psychiatric disorders
* Pregnant females
* Head trauma or injury that resulted in loss of consciousness
* MRI contraindication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-02; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Completion | 60 days
  We anticipate that participants will complete at least 30-days of the intervention.
Proximal outcomes | 60 days
  We anticipate that proximal measures of symptoms will show improvement following the training in terms of emotional reactivity, implicit emotion regulation, negative emotional memory bias, attentional bias for threat, executive functions behaviorally and N-back during fMRI as well as resting-state fMRI connectivity.
Distal outcomes | 5 months
  We anticipate that anxiety and depression symptoms, explicit emotion regulation capacities and quality of life reported on self-report measures will show improvement.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System (VAPAHCS), Palo Alto, California
  - Stanford University Department of Pscyhiatry and Behavioral Sciences, Stanford, California